CLINICAL TRIAL: NCT07194629
Title: Impact of Silver Diamine Fluoride (SDF) 38% Application on the Oral Health of the Elderly With Loss of Autonomy Living in Long-term Care Homes (CHSLDs): A Pilot and Feasibility Effectiveness Study
Brief Title: Pilot and Feasibility Study of Impact of SDF 38% Application on Oral Health of Elderly With Autonomy Loss
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Nadia Gargouri, Assistant professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CER VN 25-26-11
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Dental Caries; Elderly; Loss of Autonomy; Silver Diamine Fluoride
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Parallel-group RCT with a delayed intervention for the control group
Who Masked: Participant, Outcomes Assessor
Masking Description: The statistician will be masked as well. The expert calibrating the dentists will also be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): This arm will be provided with the intervention
  Interventions: Drug: Silver diamine Fluoride 38%
- Control (Placebo Comparator): For ethical reasons the control arm will receive treatment after the first phase of data analysis
  Interventions: Drug: placebo solution

INTERVENTIONS:
Drug: Silver diamine Fluoride 38% — SDF 38%, applied on tooth surface for arrestation of active carious lesions and prevention of development of new carious lesions
  Arms: Intervention
Drug: placebo solution — bluish liquid designed to mimic the appearance of SDF 38%
  Arms: Control

SUMMARY:
Introduction: Dental caries constitutes a major oral health problem at a global scale for the elderly population. It impacts the health system due to its high incidence and prevalence and its associated costs. The growing population of elderly experiencing a loss of autonomy is accompanied by a decline in motor functions, which affects their ability to carry out everyday tasks such as brushing their teeth. The resulting poor oral hygiene can contribute to the onset of oral diseases. Dental caries can significantly impact the quality of life of the elderly by provoking pain, chewing difficulties, tooth loss and malnutrition. Recently, Silver Diamine Fluoride (SDF) 38% has been introduced to the market as an efficient solution for promoting oral health and arresting active caries. SDF is a compound of silver, fluoride, and ammonia, which comes in the form of a bluish liquid and is applied in small amounts on active carious lesions. Despite its recent approval by Health Canada as a temporary solution for arresting active caries, few randomized controlled trials have evaluated its effectiveness on the institutionalized elderly.

Objectives: This pilot study aims to evaluate the impact of SDF on the oral health of the elderly living in long-term care facilities.

Principal objective: evaluate effectiveness of SDF on arrestation of active caries when applied for the elderly with loss of autonomy in long-term care facilities.

Secondary objectives:

1. evaluate the relationship between SDF application and caries activity
2. Analysis of salivary biomarkers involved in the associated inflammatory processes.

Methodology: A randomized controlled feasibility and effectiveness study design will be employed. This study will span over 12 months and will include 3 data collection phases.

At T0 (baseline): SDF group participants will receive an SDF application on their active caries. Control group participants will receive a 0.9% saline solution (placebo) application.

AT T1, 6 months after T0: First phase of data collection, the two groups will receive SDF application.

At T2, 12 months after T0: second phase of data collection, and for ethical reasons, the control group, who received placebo at T0, will receive an SDF application.

At the end of the project, a fluoride varnish application will be carried out on both groups to prolong preventive effects of treatment. A short questionnaire will also be shared with participants to evaluate their satisfaction and identify unintended adverse effects.

Anticipated results:

Demonstrate the efficiency of SDF in controlling active caries in the elderly with autonomy loss.

Elaborate a clinical protocol for SDF application in long-term care facilities Establish the required sample size for a future bigger study.

ELIGIBILITY:
Inclusion Criteria:

* Elderly of 65 years of age or older living at a long-term care facility targeted by the study.
* Should present at least one coronal or radicular active carious lesion that is asymptomatic, untreated, or a residual lesion under a restoration, and without pulp involvement.

Exclusion Criteria:

* Participants with inadequate collaboration that may impede dental examination or treatment.
* Participants with cardiac valve prostheses, a history of bacterial endocarditis, or valve disease following a heart transplant.
* Completely edentulous elderly, as well as elderly presenting with no coronal or radicular caries
* Participants allergic to silver, fluoride or ammonia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Arrestation of active dental caries | 0 (baseline)- 6 months (T1)- 12 months (T2)
  Evaluate the association between SDF 38% application and caries activity which will be measured at the end of the study by:
  1. Number of active carious lesions
     Description: Count of clinically active coronal or radicular carious lesions.
     Unit of measure: Number of lesions per participant.
     Measurement tool: Visual-tactile clinical examination using ICDAS II criteria.
  2. Number of carious lesions arrested by remineralization
     Description: Count of previously active lesions that present clinical signs of arrest (hard, shiny surface, absence of progression).
     Unit of measure: Number of arrested lesions per participant.
     Measurement tool: Visual-tactile clinical examination using ICDAS II criteria.
  3. Number of reactivated carious lesions (where applicable)
  Description: Count of previously arrested lesions that show new signs of activity.
  Unit of measure: Number of reactivated lesions per participant.
  Measurement tool: Visual-tactile clinical examination using ICDAS II criteria.

SECONDARY OUTCOMES:
Salivary biomarkers | 0 (baseline)- 6 months (T1)- 12 months (T2)
  Salivary biomarkers involved in remineralization of enamel and tertiary dentin and the associated inflammatory processes
Appreciation of participant | 12 months(T2)
  Elderly and their representatives' appreciation of participation in the study evaluated by questionnaire
Sample size estimation | 12 months(T2)
  Sample size estimation for a future study

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Université de Montréal, Montreal, Quebec
  - Institut universitaire de gériatrie de Montreal, Montreal, Quebec
  - CHSLD Alfred Desrochers, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sophie DOMÉJEAN , D.M., Lucas VAN DER SLUIS, Nicolas DECERLE, John DB FEATHERSTONE, Évaluation CAMBRA du risque carieux : version française. editionscdp.fr, 2012. 04
- [Background] Osterholm MT, MacDonald KL, White KE, Wells JG, Spika JS, Potter ME, Forfang JC, Sorenson RM, Milloy PT, Blake PA. An outbreak of a newly recognized chronic diarrhea syndrome associated with raw milk consumption. JAMA. 1986 Jul 25;256(4):484-90. PMID 3487659
- [Background] AlQranei MS, Balhaddad AA, Melo MAS. The burden of root caries: Updated perspectives and advances on management strategies. Gerodontology. 2021 Jun;38(2):136-153. doi: 10.1111/ger.12511. Epub 2020 Nov 24. PMID 33236462
- [Background] Gugnani N, Pandit IK, Srivastava N, Gupta M, Sharma M. International Caries Detection and Assessment System (ICDAS): A New Concept. Int J Clin Pediatr Dent. 2011 May-Aug;4(2):93-100. doi: 10.5005/jp-journals-10005-1089. Epub 2010 Apr 15. PMID 27672245
- [Background] Li R, Lo EC, Liu BY, Wong MC, Chu CH. Randomized clinical trial on arresting dental root caries through silver diammine fluoride applications in community-dwelling elders. J Dent. 2016 Aug;51:15-20. doi: 10.1016/j.jdent.2016.05.005. Epub 2016 May 18. PMID 27208876
- [Background] Siqueira GSA, Hagemann PMS, Coelho DS, Santos FHD, Bertolucci PHF. Can MoCA and MMSE Be Interchangeable Cognitive Screening Tools? A Systematic Review. Gerontologist. 2019 Nov 16;59(6):e743-e763. doi: 10.1093/geront/gny126. PMID 30517634
- [Background] Featherstone JDB, Chaffee BW. The Evidence for Caries Management by Risk Assessment (CAMBRA(R)). Adv Dent Res. 2018 Feb;29(1):9-14. doi: 10.1177/0022034517736500. PMID 29355423
- [Background] Horst JA. Silver Fluoride as a Treatment for Dental Caries. Adv Dent Res. 2018 Feb;29(1):135-140. doi: 10.1177/0022034517743750. PMID 29355428
- [Background] Santé, O.m.d.l., Prévention et traitement des caries dentaires avec des produits sans mercure et une intervention minimale : Série de notes d'information de l'OMS sur la santé buccodentaire. 2022
- [Background] Rosenblatt A, Stamford TC, Niederman R. Silver diamine fluoride: a caries "silver-fluoride bullet". J Dent Res. 2009 Feb;88(2):116-25. doi: 10.1177/0022034508329406. PMID 19278981
- [Background] Hobdell M, Petersen PE, Clarkson J, Johnson N. Global goals for oral health 2020. Int Dent J. 2003 Oct;53(5):285-8. doi: 10.1111/j.1875-595x.2003.tb00761.x. No abstract available. PMID 14560802
- [Background] Seifo N, Cassie H, Radford JR, Innes NPT. Silver diamine fluoride for managing carious lesions: an umbrella review. BMC Oral Health. 2019 Jul 12;19(1):145. doi: 10.1186/s12903-019-0830-5. PMID 31299955
- [Background] Worthington HV, Lewis SR, Glenny AM, Huang SS, Innes NP, O'Malley L, Riley P, Walsh T, Wong MCM, Clarkson JE, Veitz-Keenan A. Topical silver diamine fluoride (SDF) for preventing and managing dental caries in children and adults. Cochrane Database Syst Rev. 2024 Nov 7;11(11):CD012718. doi: 10.1002/14651858.CD012718.pub2. PMID 39508296
- [Background] Oliveira BH, Cunha-Cruz J, Rajendra A, Niederman R. Controlling caries in exposed root surfaces with silver diamine fluoride: A systematic review with meta-analysis. J Am Dent Assoc. 2018 Aug;149(8):671-679.e1. doi: 10.1016/j.adaj.2018.03.028. Epub 2018 May 24. PMID 29805039
- [Background] McReynolds D, Duane B. Systematic review finds that silver diamine fluoride is effective for both root caries prevention and arrest in older adults. Evid Based Dent. 2018 Jun;19(2):46-47. doi: 10.1038/sj.ebd.6401304. PMID 29930359
- [Background] Grandjean ML, Maccarone NR, McKenna G, Muller F, Srinivasan M. Silver Diamine Fluoride (SDF) in the management of root caries in elders: a systematic review and meta-analysis. Swiss Dent J. 2021 May 10;131(5):417-424. doi: 10.61872/sdj-2021-05-02. Epub 2021 Jan 29. PMID 33515230
- [Background] Dhanapriyanka M, Kosgallana S, Kanthi RDFC, Jayasekara P, Dao TMA, Ha DH, Do L. Professionally applied fluorides for preventing and arresting dental caries in low- and middle-income countries: Systematic review. J Public Health Dent. 2024 Jun;84(2):213-227. doi: 10.1111/jphd.12617. Epub 2024 Apr 16. PMID 38623701
- [Background] Crystal YO, Niederman R. Evidence-Based Dentistry Update on Silver Diamine Fluoride. Dent Clin North Am. 2019 Jan;63(1):45-68. doi: 10.1016/j.cden.2018.08.011. PMID 30447792
- [Background] Chan AKY, Tamrakar M, Jiang CM, Tsang YC, Leung KCM, Chu CH. Clinical evidence for professionally applied fluoride therapy to prevent and arrest dental caries in older adults: A systematic review. J Dent. 2022 Oct;125:104273. doi: 10.1016/j.jdent.2022.104273. Epub 2022 Sep 1. PMID 36058347
- [Background] Wassef, N., Utilisation du fluorure diamine d'argent en santé dentaire publique. 2019
- [Background] ENGLANDER HR, JAMES VE, MASSLER M. Histologic effects of silver nitrate of human dentin and pulp. J Am Dent Assoc. 1958 Nov;57(5):621-30. doi: 10.14219/jada.archive.1958.0258. No abstract available. PMID 13587128
- [Background] Gao SS, Zhang S, Mei ML, Lo EC, Chu CH. Caries remineralisation and arresting effect in children by professionally applied fluoride treatment - a systematic review. BMC Oral Health. 2016 Feb 1;16:12. doi: 10.1186/s12903-016-0171-6. PMID 26831727
- [Background] Hendre AD, Taylor GW, Chavez EM, Hyde S. A systematic review of silver diamine fluoride: Effectiveness and application in older adults. Gerodontology. 2017 Dec;34(4):411-419. doi: 10.1111/ger.12294. Epub 2017 Aug 15. PMID 28812312
- [Background] Association, C.D., The state of oral health in Canada. Canadian Dental Association: Ottawa, ON, Canada, 2017
- [Background] Khan A, Untoo R, Patthi B, Singla A, Kumari M, Rajeev A. Oral Health-Related Quality of Life (OHRQoL) in Elderly Patients with and without Alzheimer's Disease - An Evaluative Study. Indian J Dent Res. 2024 Apr 1;35(2):149-153. doi: 10.4103/ijdr.ijdr_792_21. Epub 2024 Sep 14. PMID 39282766
- [Background] Bellander L, Angelini E, Andersson P, Hagglin C, Wijk H. A preventive care approach for oral health in nursing homes: a qualitative study of healthcare workers' experiences. BMC Geriatr. 2024 Oct 1;24(1):803. doi: 10.1186/s12877-024-05396-1. PMID 39354356
- [Background] Yu S, Huang S, Song S, Lin J, Liu F. Impact of oral health literacy on oral health behaviors and outcomes among the older adults: a scoping review. BMC Geriatr. 2024 Oct 22;24(1):858. doi: 10.1186/s12877-024-05469-1. PMID 39438807
- [Background] Limo L, Nicholson K, Stranges S, Gomaa NA. Age and sex differences in the association of dental visits with inadequate oral health and multimorbidity: Findings from the Canadian Longitudinal Study on Aging (CLSA). BMC Public Health. 2024 Oct 25;24(1):2968. doi: 10.1186/s12889-024-20412-0. PMID 39455960
- [Background] Matthews DC, Brillant MG, Clovis JB, McNally ME, Filiaggi MJ, Kotzer RD, Lawrence HP. Assessing the oral health of an ageing population: methods, challenges and predictors of survey participation. Gerodontology. 2012 Jun;29(2):e656-66. doi: 10.1111/j.1741-2358.2011.00540.x. Epub 2011 Sep 14. PMID 21916953
- [Background] McNally ME, Martin-Misener R, Wyatt CC, McNeil KP, Crowell SJ, Matthews DC, Clovis JB. Action planning for daily mouth care in long-term care: the brushing up on mouth care project. Nurs Res Pract. 2012;2012:368356. doi: 10.1155/2012/368356. Epub 2012 Apr 5. PMID 22550572
- [Background] Jablonski RA, Munro CL, Grap MJ, Elswick RK. The role of biobehavioral, environmental, and social forces on oral health disparities in frail and functionally dependent nursing home elders. Biol Res Nurs. 2005 Jul;7(1):75-82. doi: 10.1177/1099800405275726. PMID 15920005
- [Background] https://secure.cihi.ca/free_products/Dementia_AIB_2010_EN.pdf
- [Background] Chalmers JM, Carter KD, Spencer AJ. Oral diseases and conditions in community-living older adults with and without dementia. Spec Care Dentist. 2003;23(1):7-17. doi: 10.1111/j.1754-4505.2003.tb00283.x. PMID 12887148
- [Background] Wyatt CC, So FH, Williams PM, Mithani A, Zed CM, Yen EH. The development, implementation, utilization and outcomes of a comprehensive dental program for older adults residing in long-term care facilities. J Can Dent Assoc. 2006 Jun;72(5):419. PMID 16772065
- [Background] Wyatt CC. A 5-year follow-up of older adults residing in long-term care facilities: utilisation of a comprehensive dental programme. Gerodontology. 2009 Dec;26(4):282-90. doi: 10.1111/j.1741-2358.2009.00305.x. Epub 2009 Aug 13. PMID 19682096
- [Background] Wyatt CC. Elderly Canadians residing in long-term care hospitals: Part II. Dental caries status. J Can Dent Assoc. 2002 Jun;68(6):359-63. PMID 12034072
- [Background] Wyatt CC. Elderly Canadians residing in long-term care hospitals: Part I. Medical and dental status. J Can Dent Assoc. 2002 Jun;68(6):353-8. PMID 12034071
- [Background] Woo J, Ho SC, Yu AL, Lau J. An estimate of long-term care needs and identification of risk factors for institutionalization among Hong Kong Chinese aged 70 years and over. J Gerontol A Biol Sci Med Sci. 2000 Feb;55(2):M64-9. doi: 10.1093/gerona/55.2.m64. PMID 10737687
- [Background] Sweeney MP, Williams C, Kennedy C, Macpherson LM, Turner S, Bagg J. Oral health care and status of elderly care home residents in Glasgow. Community Dent Health. 2007 Mar;24(1):37-42. PMID 17405469
- [Background] Matthews DC, Clovis JB, Brillant MG, Filiaggi MJ, McNally ME, Kotzer RD, Lawrence HP. Oral health status of long-term care residents-a vulnerable population. J Can Dent Assoc. 2012;78:c3. PMID 22364866
- [Background] Corbeil, P., J.-M. Brodeur, and S. Arpin, Étude exploratoire des problèmes de santé buccodentaire des personnes âgées hébergées en CHSLD en Montérégie, à Montréal et à Québec: rapport général. 2006: Agence de la santé et des services sociaux de la Montérégie.
- [Background] van der Maarel-Wierink CD, Vanobbergen JN, Bronkhorst EM, Schols JM, de Baat C. Risk factors for aspiration pneumonia in frail older people: a systematic literature review. J Am Med Dir Assoc. 2011 Jun;12(5):344-54. doi: 10.1016/j.jamda.2010.12.099. Epub 2011 Mar 21. PMID 21450240
- [Background] Taylor GW, Loesche WJ, Terpenning MS. Impact of oral diseases on systemic health in the elderly: diabetes mellitus and aspiration pneumonia. J Public Health Dent. 2000 Fall;60(4):313-20. doi: 10.1111/j.1752-7325.2000.tb03341.x. PMID 11243053
- [Background] Sjogren P, Nilsson E, Forsell M, Johansson O, Hoogstraate J. A systematic review of the preventive effect of oral hygiene on pneumonia and respiratory tract infection in elderly people in hospitals and nursing homes: effect estimates and methodological quality of randomized controlled trials. J Am Geriatr Soc. 2008 Nov;56(11):2124-30. doi: 10.1111/j.1532-5415.2008.01926.x. Epub 2008 Sep 15. PMID 18795989
- [Background] Quagliarello V, Juthani-Mehta M, Ginter S, Towle V, Allore H, Tinetti M. Pilot testing of intervention protocols to prevent pneumonia in nursing home residents. J Am Geriatr Soc. 2009 Jul;57(7):1226-31. doi: 10.1111/j.1532-5415.2009.02311.x. Epub 2009 Jun 3. PMID 19558483
- [Background] Muller F. Oral hygiene reduces the mortality from aspiration pneumonia in frail elders. J Dent Res. 2015 Mar;94(3 Suppl):14S-16S. doi: 10.1177/0022034514552494. Epub 2014 Oct 7. No abstract available. PMID 25294365
- [Background] Montebugnoli L, Servidio D, Miaton RA, Prati C, Tricoci P, Melloni C. Poor oral health is associated with coronary heart disease and elevated systemic inflammatory and haemostatic factors. J Clin Periodontol. 2004 Jan;31(1):25-9. doi: 10.1111/j.0303-6979.2004.00432.x. PMID 15058371
- [Background] El-Solh AA. Association between pneumonia and oral care in nursing home residents. Lung. 2011 Jun;189(3):173-80. doi: 10.1007/s00408-011-9297-0. Epub 2011 Apr 30. PMID 21533635
- [Background] Beck JD, Offenbacher S. Oral health and systemic disease: periodontitis and cardiovascular disease. J Dent Educ. 1998 Oct;62(10):859-70. No abstract available. PMID 9847889
- [Background] Bassim CW, Gibson G, Ward T, Paphides BM, Denucci DJ. Modification of the risk of mortality from pneumonia with oral hygiene care. J Am Geriatr Soc. 2008 Sep;56(9):1601-7. doi: 10.1111/j.1532-5415.2008.01825.x. Epub 2008 Aug 4. PMID 18691286
- [Background] Azarpazhooh A, Leake JL. Systematic review of the association between respiratory diseases and oral health. J Periodontol. 2006 Sep;77(9):1465-82. doi: 10.1902/jop.2006.060010. PMID 16945022
- [Background] Hopcraft MS, Morgan MV, Satur JG, Wright FA. Edentulism and dental caries in Victorian nursing homes. Gerodontology. 2012 Jun;29(2):e512-9. doi: 10.1111/j.1741-2358.2011.00510.x. Epub 2011 Jun 28. PMID 21707743
- [Background] Zuluaga DJ, Ferreira J, Montoya JA, Willumsen T. Oral health in institutionalised elderly people in Oslo, Norway and its relationship with dependence and cognitive impairment. Gerodontology. 2012 Jun;29(2):e420-6. doi: 10.1111/j.1741-2358.2011.00490.x. Epub 2011 May 12. PMID 21564272
- [Background] Silva M, Hopcraft M, Morgan M. Dental caries in Victorian nursing homes. Aust Dent J. 2014 Sep;59(3):321-8. doi: 10.1111/adj.12188. Epub 2014 Jul 22. PMID 24819713
- [Background] Petelin M, Cotic J, Perkic K, Pavlic A. Oral health of the elderly living in residential homes in Slovenia. Gerodontology. 2012 Jun;29(2):e447-57. doi: 10.1111/j.1741-2358.2011.00497.x. Epub 2011 May 25. PMID 21615469
- [Background] Laurent M, Gogly B, Tahmasebi F, Paillaud E. [Oropharyngeal candidiasis in elderly patients]. Geriatr Psychol Neuropsychiatr Vieil. 2011 Mar;9(1):21-8. doi: 10.1684/pnv.2011.0259. French. PMID 21586373
- [Background] Lamy M. [Bucco-dental health in the elderly]. Rev Med Liege. 2014 May-Jun;69(5-6):357-60. French. PMID 25065245
- [Background] https://statistique.quebec.ca/fr/fichier/bilan-demographique-quebec-edition-2023.pdf
- [Background] Hopcraft MS, Morgan MV, Satur JG, Wright FA, Darby IB. Oral hygiene and periodontal disease in Victorian nursing homes. Gerodontology. 2012 Jun;29(2):e220-8. doi: 10.1111/j.1741-2358.2010.00448.x. Epub 2010 Nov 17. PMID 21083744
- [Background] Chen X, Clark JJ, Naorungroj S. Oral health in nursing home residents with different cognitive statuses. Gerodontology. 2013 Mar;30(1):49-60. doi: 10.1111/j.1741-2358.2012.00644.x. Epub 2012 Feb 26. PMID 22364512
- [Background] Chalmers J, Pearson A. Oral hygiene care for residents with dementia: a literature review. J Adv Nurs. 2005 Nov;52(4):410-9. doi: 10.1111/j.1365-2648.2005.03605.x. PMID 16268845
- [Background] https://statistique.quebec.ca/fr/fichier/bilan-demographique-quebec-edition-2024.pdf
- [Background] https://statistique.quebec.ca/fr/fichier/perspectives-demographiques-quebec-et-regions-2021-2071-edition-2024.pdf
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of untreated caries: a systematic review and metaregression. J Dent Res. 2015 May;94(5):650-8. doi: 10.1177/0022034515573272. Epub 2015 Mar 4. PMID 25740856
- See also: Related Info — https://statistique.quebec.ca/fr/fichier/bilan-demographique-quebec-edition-2023.pdf